CLINICAL TRIAL: NCT06896253
Title: Pulse Corticosteroids Or/and Immunoglobulins to Treat Fulminant Myocarditis: a Double-blind Randomized Controlled Adaptive Trial the CORIUM Study
Brief Title: Pulse Corticosteroids Or/and Immunoglobulins to Treat Fulminant Myocarditis
Acronym: CORIUM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP220808; 2023-506599-28-01 (EU CTIS Number)
Record Dates: First submitted 2025-02-12; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Myocarditis Acute
Keywords: Fulminant myocarditis
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pulse bolus corticosteroids group (Experimental): 1. 1 gram/day of methylprednisolone IV for three days followed by 1mg/kg/day IV until inotropes weaning or 7 days whatever come first.
  2. Placebo of IVIG: glucose 5% 0.5g/kg/day for 4 days
  Interventions: Drug: Pulse bolus corticosteroids
- Pulse bolus corticosteroids and IVIG group (Experimental): 1. 1 gram/day of methylprednisolone IV for three days followed by 1mg/kg/day IV until inotropes weaning or 7 days whatever come first.
  2. 0.5g/kg/day IVIG for 4 days.
  Interventions: Drug: Pulse bolus corticosteroids and IVIG
- Double placebo pulse bolus corticosteroids (G5%) and IVIG (G5 %) (Placebo Comparator)
  Interventions: Drug: Pulse bolus corticosteroids (G5%) and IVIG (G5 %)

INTERVENTIONS:
Drug: Pulse bolus corticosteroids — Treatment administration
  Arms: Pulse bolus corticosteroids group
Drug: Pulse bolus corticosteroids and IVIG — Treatment administration
  Arms: Pulse bolus corticosteroids and IVIG group
Drug: Pulse bolus corticosteroids (G5%) and IVIG (G5 %) — Treatment administration
  Arms: Double placebo pulse bolus corticosteroids (G5%) and IVIG (G5 %)

SUMMARY:
Fulminant myocarditis (FM) is the most severe manifestation of acute myocarditis, an acute inflammatory myocardial disease most often triggered by viral infections.

Currently, the most accepted definition of FM requires acute illness, hemodynamic compromise due to cardiogenic shock, and need for hemodynamic support (inotropes and/or temporary mechanical circulatory support (t-MCS) in the absence of an ischemic cause or other pre-existing cardiomyopathies. Unfortunately, there is a paucity of evidence-based management strategies for this disease and the management of patients affected by FM often varies according to local experience and practice with the role of immunosuppression being the most debated issue.

Besides, due to inconsistent results obtained in several studies and frequent spontaneous recovery with supportive therapy alone, immunosuppression is largely debated in the setting of lymphocytic myocarditis (LM). Among available medications for this disease, corticosteroids are often used despite a lack of clear evidence in the context of FM. Similarly, intravenous immunoglobulin (IVIG) has both antiviral and anti-inflammatory effects on myocarditis. In adults, a recent meta-analysis based on case series showed that IVIG therapy significantly reduced in-hospital mortality, improved the left ventricular ejection fraction, and significantly increased the survival rate in patients with FM. More recently, FM among patients with COVID-19, including post-infectious multisystem inflammatory syndrome, has been reported in young adult patients. These severe forms have been successfully treated with intravenous corticosteroids and IVIG, highlighting the relevance of the systemic inflammatory response in determining cardiac injury in COVID-19, even though more evidence is needed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Fulminant myocarditis defined by

  * the acute illness (<1 month from symptom onset),
  * hemodynamic compromise due to cardiogenic shock (confirmed by echocardiography) or electrical storm,
  * elevated plasma cardiac troponin > twice normal value
  * need for hemodynamic support (inotropes or temporary mechanical circulatory support) for less than 72 hours in the absence of an ischemic cause or other pre-existing cardiomyopathies Noticeably, a coronary angiogram should be performed in patients ≥40 years of age when myocarditis has not been proven histologically. Besides, an endomyocardial biopsy will not be mandatory to fulfill the definition of fulminant myocarditis.

    2. Signed informed consent from the patient, a close relative or surrogate or a family member or a legal representative for minor patient.
  * Adult : According to the specifications of emergency inclusion, randomization without the close relative/surrogate consent could be performed if the patientis unable to give his/her consent and when the close relative/surrogate/family member are absent. Close relative/surrogate/family member consent will be asked as soon as possible after randomization. The patient will be asked as soon as possible to give his/her consent for the continuation of the trial when his/her condition will allow.
  * Minor : According to the specifications of emergency inclusion, randomization could be performed when legal representative are absent. Legal representative consent will be asked as soon as possible after randomization 3. Social security registration (AME excluded)

Exclusion Criteria:

* 1. Age <15 2. Pregnancy or breastfeeding or baby delivery <6 months 3. Initiation of inotropes or temporary mechanical circulatory support >72 hours 4. Resuscitation >20 minutes (cumulative low-flow time > 20 minutes ) 5. Pre-existing ischemic or dilated cardiomyopathy or Tako-Tsubo evaluated by echocardiography.

  6. Known systemic autoimmune disorder or other conditions requiring immunosuppression 7. Patients with peripheral eosinophilia (≥1000 G/L) 8. Myocarditis associated with anti-cancer immune checkpoint inhibitor agents 9. Active severe bacterial or fungal infectious disease 10. Patient moribund on the day of randomization, SAPS II >90 11. Contraindication or allergies to corticosteroids or immunoglobulins or any components of the formulations or their excipients 12. Patients already on corticosteroids or receiving IVIG 13. Participation in another interventional study or being in the exclusion period at the end of a previous study.

  14. Patients with an uncontrolled psychotic condition Patients with known anti-IgA antibodies in line with the contraindications of methylprednisolone IV and of IVIg based products respectively

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
A composite hierarchical outcome composed of four components : 1) mortality at D28 2) heart transplant/VAD/persisting t-MCS at D28, and 3) number of days alive without t-MCS and inotropes at D28 | Day 28
  Each patient will be compared with every other patient in the study and assigned a score (tie: 0, win: +1, loss: -1) for each pairwise comparison based on whom fared better. If one patient survived without heart transplantation or long-term assist ventricular device or t-MCS still ongoing at day 28 and the other does not, scores of +1 and -1 will be assigned, respectively. Otherwise, the assigned score will depend on which patient had more days free from t-MCS and inotropes: the patient with more days off t-MCS and inotropes will receive a score of +1, and the other patient -1. If both patients survived and had the same number of days off t-MCS and inotropes, or if both patients died or had a heart transplant or a VAD, they will be both assigned a score of 0 for that pairwise comparison. For each patient, scores for all pairwise comparisons will be summed, resulting in a cumulative score which will be the primary endpoint of the study.

SECONDARY OUTCOMES:
Mortality | Day 28, Day 60, Day 90
Number of temporary mechanical circulatory support free days | Day 28
Number of inotropes-free days | Day 28
Incidence of ventricular assisted device use | Day 28, Day 60, Day 90
Incidence of heart transplant | Day 28, Day 60, Day 90
Left ventricular function (%) assessed by echocardiography (Simpson method) | Day 3, Day 7, Day 14, Day 28
Time to normalize troponin | From randomization to Day 14
Time to normalize N-terminal pro-B-type natriuretic peptide | From randomization to Day 14
Incidence of drugs side effects | From randomization to Day 28
  nosocomial infections, significant gastrointestinal bleeding, renal insufficiency, acute delirium leading to the use of neuroleptic agents
Proportion of patients with left ventricular ejection fraction < 55% | Day 28, 6 months
Proportion of patients with left ventricular dilatation | Day 28, 6 months
Proportion of patients with late gadolinium enhancement evaluated by cardiac magnetic resonance imaging | 6 months
Incidence of hyperglycemia | From randomization to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Alain COMBES, MD, Study Director — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal